CLINICAL TRIAL: NCT01401257
Title: A Phase II, Randomized, Placebo-controlled Trial of the Safety, Efficacy, Pharmacodynamics and Pharmacokinetics of PXT3003 in Patients With Charcot-Marie-Tooth Disease Type 1A.
Brief Title: Phase II, Randomized, Placebo-controlled Trial in Patients With Charcot-marie-tooth Disease Type 1A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharnext S.C.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLN-PXT3003-01
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Charcot-Marie-Tooth Disease; Hereditary Neuropathy With Liability to Pressure Palsies; Genetic Disorders
Keywords: PXT3003; Charcot-Marie-Tooth Disease; Hereditary Motor and Sensory Neuropathies
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Tomaculous neuropathy; Genetic Diseases, Inborn; Hereditary Sensory and Motor Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PXT3003 Low dose (Experimental): Oral Liquid formulation, 1/100, bid, 12 months
  Interventions: Drug: PXT3003 Low dose
- PXT3003 Intermediate dose (Experimental): Oral Liquid formulation, 1/50, bid, 12 months
  Interventions: Drug: PXT3003 Intermediate Dose
- PXT3003 High dose (Experimental): Oral Liquid formulation, 1/10, bid, 12 months
  Interventions: Drug: PXT3003 High Dose
- Placebo (Placebo Comparator): Oral Liquid formulation, bid, 12 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PXT3003 Low dose — Liquid,5 ml, twice a day, 12-month treatment
  Other Names: Pleocompound PXT3003
  Arms: PXT3003 Low dose
Drug: PXT3003 Intermediate Dose — Liquid,5 ml, twice a day, 12-month treatment
  Other Names: Pleocompound PXT3003
  Arms: PXT3003 Intermediate dose
Drug: PXT3003 High Dose — Liquid,5 ml, twice a day, 12-month treatment
  Other Names: Pleocompound PXT3003
  Arms: PXT3003 High dose
Other: Placebo — Liquid,5 ml, twice a day, 12-month treatment
  Other Names: Pleocompound PXT3003
  Arms: Placebo

SUMMARY:
The present trial is a randomized, placebo-controlled study evaluating 3 different doses of PXT3003 in patients with CMT1A disease.

DETAILED DESCRIPTION:
In addition to the safety and tolerability of the treatment, clinical, electrophysiological and biological endpoints (PMP22 mRNA, skin biopsy histology and plasma biomarkers) will be assessed. Standard laboratory tests and drug plasma concentrations will also be measured. Because of the slow progression of the disease and the nature of the observed symptoms, a minimum duration of 12 months of treatment is required in order to observe a potential improvement in any of the efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

* DNA proven CMT1A
* Muscle weakness in at least foot dorsiflexion (clinical assessment)
* Age between 18 and 65 years
* Male or non pregnant, non breastfeeding female
* CMT neuropathy score at screening ≤ 20
* Agrees to perform electrorophysiological studies and two cutaneous biopsies for determination of PMP22 expression and histology
* Providing signed written informed consent to participate in the study and willing and able to comply with all study procedures and scheduled visits

Exclusion Criteria:

* Patients with another neurological disease
* Patients using unauthorized concomitant treatments, ascorbic acid, opioids, levothyroxine and potentially neurotoxic drugs. Patients who can/agree to stop these medications 4 weeks before randomization can be included
* Patients who have participated in another trial of investigational drug within the past 30 days
* Concomitant major systemic disease
* Clinically significant history of unstable medical illness over the last 30 days (unstable angina…)
* History of significant hematologic, kidney, liver disease, or insulin-dependent diabetes
* Clinically significant abnormalities on the prestudy laboratory evaluation, physical evaluation, electrocardiogram (ECG)
* ASAT/ALAT levels above the upper limit of normal (ULN). However, patients with an isolated elevation of either ASAT or ALAT (<1.5 ULN) can be included at investigators" discretion if the remaining liver function tests are normal and if ASAT or ALAT value is stable at 2 distinct evaluations in the month prior to inclusion
* Serum creatinine levels above the upper limit of normal
* Limited mental capacity or psychiatric disease rendering the subject unable to provide written informed consent or comply with evaluation procedures
* History of recent alcohol or drug abuse or non-adherence with treatment or other experimental protocols
* Female of childbearing potential (apart of patient using adequate contraceptive measures), pregnant or breast feeding
* Suspected inability to complete the study follow-up (foreign workers, transient visitors, tourists or any others for whom follow-up evaluation is not assured)
* Limb surgery in the six months before randomization or planned before completion of the trial
* Known hypersensitivity to any of the individual components of PXT3003
* Porphyria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahram ATTARIAN, MD, Principal Investigator — Hôpital La Timone; Viviane BERTRAND, PhD, Study Director — Pharnext S.C.A.
Locations (6):
- France (6):
  - Hôpital Roger Salengro, Lille
  - CHU Dupuytren, Limoges
  - CHU Lyon Sud, Lyon
  - Hôpital La Timone, Marseille
  - Hôtel Dieu, Nantes
  - Groupe Hospitalier Pitié-Salpétrière, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Attarian S, Vallat JM, Magy L, Funalot B, Gonnaud PM, Lacour A, Pereon Y, Dubourg O, Pouget J, Micallef J, Franques J, Lefebvre MN, Ghorab K, Al-Moussawi M, Tiffreau V, Preudhomme M, Magot A, Leclair-Visonneau L, Stojkovic T, Bossi L, Lehert P, Gilbert W, Bertrand V, Mandel J, Milet A, Hajj R, Boudiaf L, Scart-Gres C, Nabirotchkin S, Guedj M, Chumakov I, Cohen D. An exploratory randomised double-blind and placebo-controlled phase 2 study of a combination of baclofen, naltrexone and sorbitol (PXT3003) in patients with Charcot-Marie-Tooth disease type 1A. Orphanet J Rare Dis. 2014 Dec 18;9:199. doi: 10.1186/s13023-014-0199-0. PMID 25519680

RESULTS

PARTICIPANT FLOW:
Groups:
- PXT3003 Low Dose: Oral Liquid formulation, 1/100, bid, 12 months
  PXT3003: Liquid,5 ml, twice a day, 12-month treatment
- PXT3003 Intermediate Dose: Oral Liquid formulation, 1/50, bid, 12 months
  PXT3003: Liquid,5 ml, twice a day, 12-month treatment
- PXT3003 High Dose: Oral Liquid formulation, 1/10, bid, 12 months
  PXT3003: Liquid,5 ml, twice a day, 12-month treatment
Period: Overall Study
Arm/Group | PXT3003 Low Dose | PXT3003 Intermediate Dose | PXT3003 High Dose | Placebo
Started | 21 | 21 | 19 | 19
Completed | 21 | 19 | 16 | 17
Not Completed | 0 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PXT3003 Low Dose | PXT3003 Intermediate Dose | PXT3003 High Dose | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 19 | 19 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 19 | 19 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 47.9 [18 to 63] | 44.3 [23 to 64] | 44.6 [24 to 63] | 43.2 [21 to 65] | 45.1 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 10 | 11 | 48
  Male | 7 | 8 | 9 | 8 | 32
Region of Enrollment [Number; unit: participants]
  France | 21 | 21 | 19 | 19 | 80

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of PXT3003
Description: The Primary Objective is to assess the clinical and laboratory safety and tolerability of three doses of PXT3003 administered orally for 12 months to CMT1A patients versus placebo.
  Number of participants with adverse events in each arm.
Time Frame: Screening, randomization, 1-, 3-, 6-, 9-, 12-month treatment and 1-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | PXT3003 Low Dose | PXT3003 Intermediate Dose | PXT3003 High Dose | Placebo
Number analyzed (Participants) | 21 | 21 | 19 | 19
Participants | 21 | 21 | 19 | 19

2. Secondary Outcome: To Obtain Preliminary Data on the Efficacy of PXT3003 on Clinical Scores and Functional Tests
Description: Efficacy scores and functional tests will be assessed CMTNS/CMTES:ONLS, VAS, fatigue, pain, six minute walk test (6MWT), nine-hole peg test, quantified muscular testing (QMT; hand grip and foot dorsiflexion), CGI.
  For each test or score, change from baseline after 3-,6-, 9- and 12-months of treatment.
Time Frame: Screening, randomization, 3-, 6-, 9- and 12-months treatment
Reporting Status: Not Posted

3. Secondary Outcome: To Assess the Pharmacodynamic Effect of PXT3003 on PMP22 mRNA Levels and Intra-epidermal Axon Density in Cutaneous Biopsy
Description: A cutaneous biopsy (consisting in 2 small punch biopsies) will be performed to assess PMP22 mRNA expression and intra-epidermal axon density.
  Change from baseline after 12-month of treatment.
Time Frame: Randomization and 12-month treatment
Reporting Status: Not Posted

4. Secondary Outcome: To Assess the Pharmacodynamic Effect of PXT3003 on Selected Neurophysiological Parameters
Description: Electrophysiological examination will be performed to assess sensory and motor responses of the median and ulnar nerves (non-dominant side) including: NCV, compound muscle action potential (CMAP) and SNAP.
  Change from baseline after 3-,6-, 9- and 12-months of treatment.
Time Frame: Screening, randomization, 3-, 6-, 9- and 12-month treatment
Reporting Status: Not Posted

5. Secondary Outcome: To Assess the Pharmacodynamic Effect of PXT3003 on a Series of Biochemical Biomarkers
Description: Dosages of biochemical biomarkers in plasma.
  Change from baseline after 3-month of treatment.
Time Frame: Randomization and 3-month treatment
Reporting Status: Not Posted

6. Secondary Outcome: To Assess the Plasma Concentrations of PXT3003
Description: PXT3003 plasmatic concentrations after one administration (randomization) and after 1-,6-and 12-months of treatment.
Time Frame: Randomization, 1-, 6- and 12-month treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | PXT3003 Low Dose | PXT3003 Intermediate Dose | PXT3003 High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/21 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 12/21 | 10/21 | 13/19 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PXT3003 Low Dose (N=21) | PXT3003 Intermediate Dose (N=21) | PXT3003 High Dose (N=19) | Placebo (N=19)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — Unrelated to study medication
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Unrelated to study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PXT3003 Low Dose (N=21) | PXT3003 Intermediate Dose (N=21) | PXT3003 High Dose (N=19) | Placebo (N=19)
Infections and infestations (Infections and infestations) | 11 | 10 | 11 | 8
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 12 | 8 | 13 | 7
Nervous system disorders (Nervous system disorders) | 8 | 8 | 11 | 9
Gastrointestinal disorders (Gastrointestinal disorders) | 7 | 5 | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual publication (paper, abstract, poster, oral presentation) is allowed until results of the complete study have been published.

The Investigator agrees that any proposed publication, presentation or use of results arising from the Investigation will be submitted to Pharnext for review and written agreement prior to submission.